CLINICAL TRIAL: NCT03251768
Title: Efficacy and Safety Phase IIb Study of Recombinant Human Serum Albumin/ Granulocyte Colony-Stimulating Factor Fusion Protein for Injection to Prevent Neutrophilic Granulocytopenia Among Chemotherapy Breast Cancer Patients
Brief Title: Recombinant Human Serum Albumin/Granulocyte Colony Stimulating Factor Fusion Protein for Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin SinoBiotech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHS01N-1892
Record Dates: First submitted 2017-08-07; First posted 2017-08-16 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2018-12

CONDITIONS: Chemotherapy-induced Neutropenia
Keywords: Chemotherapy; Neutropenia; breast cancer
MeSH Terms: conditions — Neutropenia; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): intervention: rHSA-GCSF 2.4 mg Drug: TE or TEC TE: Taxotere+Epirubicin Taxotere (75mg/m2)and Epirubicin(75mg/m2), IV on day 1 of each 21 chemotherapy cycle.
  TEC:Taxotere+Epirubicin+Cyclophosphamide Taxotere (75mg/m2),Epirubicin (75mg/m2) and Cyclophosphamide (500mg/m2), IV on day 1 of each 21 chemotherapy cycle.
  Recombinant Human Serum Albumin/Granulocyte Colony-Stimulating Factor Fusion Protein（2.4mg）will be injected subcutaneously at at 10 am (±90 min) on the 3th and 7th day of each chemotherapy cycle.After injection, stop administrating if Absolute Neutrophil Count (ANC) in peripheral blood exceeded 5.0×109/L at two contiguous times at least. If not up to standard, investigator should decide whether or not the third administration.
  Interventions: Drug: rHSA-GCSF 2.4mg
- Positive control group (Active Comparator): intervention: GCSF Drug: TE or TEC TE: Taxotere+Epirubicin Taxotere (75mg/m2)and Epirubicin(75mg/m2), IV on day 1 of each 21 chemotherapy cycle.
  TEC:Taxotere+Epirubicin+Cyclophosphamide Taxotere (75mg/m2),Epirubicin (75mg/m2) and Cyclophosphamide (500mg/m2), IV on day 1 of each 21 chemotherapy cycle.
  Recombinant Human Granulocyte Colony-Stimulating Factor Injection (5μg/kg/day) will be injected subcutaneously at 10 am (±90 min) from the 3rd of per chemotherapy cycle. After the injection, stop administrating if Absolute Neutrophil Count (ANC) in peripheral blood exceeded 5.0×109/L at two contiguous times at least. (The minimum of usage was continuous 7 days ,The maximum of usage was continuous 14 days)
  Interventions: Drug: GCSF

INTERVENTIONS:
Drug: rHSA-GCSF 2.4mg — Human Serum Albumin GCSF 2.4mg at day 3 and day 7
  Other Names: Human Serum Albumin GCSF
  Arms: Test group
Drug: GCSF — GCSF 5 mcg/kg/day
  Other Names: jisaixin
  Arms: Positive control group

SUMMARY:
Evaluation of the efficacy and safety of recombinant human serum albumin / granulocyte-stimulating factor fusion protein for injection to prevent chemotherapy-induced neutropenia

DETAILED DESCRIPTION:
* Brief Protocol: Treat the patients taking Taxotere+Epirubicin +Cyclophosphamide (TEC) treatment or Taxotere+Epirubicin (TE)treatment chemotherapy with the study medicine or positive control during the period between two chemotherapy treatments.
* Targeted patients: breast cancer
* Subjects were randomly divided into two groups. The test group received recombinant human serum albumin / granulocyte thorns for injection Stimulant fusion protein 2.4mg treatment. Positive control group received recombinant human granulocyte colony stimuli Factor injection therapy
* Number of patients: 80

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65.
* Diagnosed breast cancer, suitable for TEC or TE .
* ECOG performance status 0 or 1.
* Adjuvant chemotherapy; new adjuvant chemotherapy; newly diagnosed class Ⅳ and prior chemotherapy.
* No obvious abnormal ecg examination.
* TBIL, ALT, AST≤2.5×ULN (≤5×ULN if presence of hepatic metastases).
* Cr, BUN≤2.5×ULN.
* Signed informed consent.

Exclusion Criteria:

* Chemotherapy within past 4 weeks.
* Uncontrolled inflammatory disease,axillary temperature≥38℃.
* Merging other malignant tumor.
* Pregnancy or nursing status.
* Participation in another clinical trial with and investigational product within 3 months prior to study entry.
* Severe diabetes mellitus, or poor blood sugar controller.
* Allergic disease or allergic constitution. History of protein allergy.
* History of drug addiction and alcoholism.
* Hematopoietic stem cell transplantation or organ transplantation.
* Antibiotics were treated within 72 hours before chemotherapy.
* Long-term use of hormones or immunosuppressive agents.
* Severe mental or neurological disease.
* Chronic disease of severe cardiac, kidney and liver.
* Other conditions that would be excluded from this study according to doctors'judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Main curative effect evaluation index | 4 weeks
  The duration of the degree of Ⅳ neutropenia

SECONDARY OUTCOMES:
Secondary efficacy evaluation index | 8 weeks
  The duration of the degree of Ⅳ neutropenia(ANC<0.5×109/L)
Secondary efficacy evaluation index-1 | 8 weeks
  The time required for neutrophil recovery to 2.0x109/L(
Secondary efficacy evaluation index-2 | 8 weeks
  ANC
Secondary efficacy evaluation index-3 | 8 weeks
  febrile neutropenia
Secondary efficacy evaluation index-4 | 8 weeks
  The usage of antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Binghe XU, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chen S, Han Y, Ouyang Q, Lu J, Zhang Q, Yang S, Wang J, Huang H, Liu H, Shao Z, Li H, Chen Z, Sun S, Geng C, Lu J, Sun J, Wang J, Xu B. Randomized and dose-escalation trials of recombinant human serum albumin /granulocyte colony-stimulating factor in patients with breast cancer receiving anthracycline-containing chemotherapy. BMC Cancer. 2021 Mar 31;21(1):341. doi: 10.1186/s12885-021-08093-z. PMID 33789616